CLINICAL TRIAL: NCT02892786
Title: Detection in Peripheral Blood of Circulating Tumor Cells in Patient With Head and Neck Squamous Cell Carcinoma
Acronym: CTCVADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-A00586-33
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Head and Neck Cancer
Keywords: circulating tumor cell; CellSearch™ method; RT-PCR
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental (Experimental)
  Interventions: Other: Circulating Tumor Cells

INTERVENTIONS:
Other: Circulating Tumor Cells — Patients with stage III and IV head and neck squamous cell carcinoma undergoing surgery were enrolled in this study
  5 and 7.5 ml of peripheral venous blood will be taken before the surgery, just at the end of surgery and one week after surgery
  Analysis was performed by RT-PCR and the CellSearch™ method using immunomagnetic and fluorescence approaches.
  Patients will be followed every 3 months for two years.

SUMMARY:
The dissemination of individual tumor cells is a common phenomenon in solid cancers. Detection of tumor cells in peripheral blood circulating tumor cells (CTC) in nonmetastatic situation is of high prognostic significance.

The objective of our study was to detect circulating tumor cells in two different method in patient with head and neck squamous cell carcinoma .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with head and neck squamous cell cancer stage III or IV histologically proven
* Patient naive to any prior therapy
* Patient with operate cancer and resectable tumor
* Hemoglobin ≥ 10g / dL
* Performance status ≤ 2
* Ability to provide written informed consent
* Patient's legal capacity to consent to study participation

Exclusion Criteria:

* Other previous histology tumors
* Medical conditions or acute or chronic severe psychiatric disorders
* Deprived of liberty or under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Circulating tumor cells in peripheral blood during head and neck surgery | 7 days
  The number of circulating tumor cells detected per milliliter of peripheral blood will be evaluated on the day before, the day of surgery and 7 days after the surgery.

SECONDARY OUTCOMES:
Comparison between RT-PCR and CellSearch™ method | 1 day
  The comparison between RT-PCR and CellSearch™ method will be the positivity sample rate
Prognostic marker of relapse | 2 years
  Local recurrence, regional or metastatic head and neck cancer in the two years

CONTACTS AND LOCATIONS:
Overall Officials: MASTRONICOLA Romina, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No